CLINICAL TRIAL: NCT05119309
Title: Monoclonal Gammopathies of Renal Significance: Clinical-histological Features of a Multicenter Case Series (MGRS Project)
Brief Title: MGRS: Clinical-histological Features of a Multicenter Case Series
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: MGRS
Record Dates: First submitted 2021-07-29; First posted 2021-11-15 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Monoclonal Gammopathy of Renal Significance
Keywords: MGRS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: Renal biopsy diagnosis of MGRS or disease linked to multiple myeloma and B cell lymphoma
- control patient group: Renal biopsy diagnosis of nephropathy linked to onco-haematological pathology with full clinical expression (Multiple Myeloma, B-cell Lymphoma)

SUMMARY:
The term "Monoclonal Gammopathies of Renal Significance" (MGRS) describes a group of diseases characterized by the presence of an immunoglobulin or monoclonal immunoglobulin fraction that has the ability to cause renal damage.

It is important to diagnose MGRS correctly and early as renal survival depends on the renal function present at the time of diagnosis and it is necessary to establish a specific treatment that aims to stop the progression of the damage. organ and restoration of renal function.

To date, there are no targeted therapeutic strategies that can prevent the formation of deposits or that can eliminate the deposits already present in the kidney, which constitute the etiopathogenetic factor of these pathologies. Therefore, the only valid therapeutic option is to act against the clone of B lymphocytes underlying the nephrological pathology, although it is not a clone with such requirements to be able to define it as a tumor.

Therefore, given the absence of a well-defined policy in the therapy of MGRS and the doubts present on the validity of a therapeutic approach aimed at the suppression of a plasma cell clone, the investigators decided to carry out an observational retrospective study with the aim of describing, in a large series of MGRS treated with oncohematological therapy, the renal and overall outcome of patients and identify any presenting prognostic characteristics that can help improve the diagnosis of these disorders and the long-term survival of patients.

DETAILED DESCRIPTION:
The group will be compared with patients suffering from renal disease associated with oncohematological diseases with full clinical expression (multiple myeloma and B cell lymphomas) which produce monoclonal component and who have been treated according to the established specific schemes of each disease.

The study will have a total duration of 12 months. It will analyze the data of the patients included in the clinical charts from 01/01/2010 to 31/12/2020. A total of 120 patients and 60 pathological controls will be enrolled (2:1 ratio), expected total number of patients from the centers participating in the study enrolled through the outpatient clinics of the Departments of the study.

The variables considered in the study are routine laboratory data (renal function, electrophoresis of serum and urinary proteins with immunofission, serum free light chains and their ratio, proteinuria 24 h serum albumin), clinical and anamnestic data, data on current drug therapy and description of renal biopsy characteristics using a predefined database with statistical analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* Renal biopsy diagnosis of MGRS or disease linked to multiple myeloma and B cell lymphoma between 01/01/2010 and 31/12/2020 (for patient group)
* Renal biopsy diagnosis of nephropathy linked to onco-haematological pathology with full clinical expression (eg Multiple Myeloma, B-cell Lymphoma) between 01/01/2010 and 31/12/2021 (for control group);
* Age greater than or equal to 18 years;
* Informed consent freely granted and acquired before the start of the study.

Exclusion Criteria:

* Patients who do not meet the relevant inclusion criteria and who do not have an established diagnosis of MGRS or disease related to multiple myeloma and B-cell lymphoma will be excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a large series of patients with Monoclonal Gammopathies of Renal Significance treated with oncohematological therapy; this group will be compared with patients suffering from renal disease associated with oncohematological diseases with full clinical expression (multiple myeloma and B cell lymphomas) which produce monoclonal component and who have been treated according to the established specific schemes of each disease.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Assessment of pictures of biochemical presentation | through study completion, an average of 1 year
  Multicenter retrospective evaluation of biochemical presentation pictures of patients with MGRS and clinically expressed haematological diseases, with renal involvement

SECONDARY OUTCOMES:
Evaluation of the renal status of study patients using physiological parameters (use of the eGFR in ml / min / 1.73 m2 calculated with CKD-EPI) | through study completion, an average of 1 year
  Renal and global health outcomes of patients with MGRS, comparison with patients with haematological diseases
Evaluation of the global health of study patients using physiological parameters (use of the eGFR in ml / min / 1.73 m2 calculated with CKD-EPI) | through study completion, an average of 1 year
  Renal and global health outcomes of patients with MGRS, comparison with patients with haematological diseases
Prognostic characteristics | through study completion, an average of 1 year
  Identification of any prognostic characteristics of presentation
Biochemical indicators of response to treatment | through study completion, an average of 1 year
  Identification of any biochemical indicators of response to treatment (serum and urinary protein electrophoresis and 24 h proteinuria to evaluate renal function)
Clinical indicators of response to treatment | through study completion, an average of 1 year
  Identification of any biochemical and clinical indicators of response to treatment (serum and urinary protein electrophoresis and 24 h proteinuria to evaluate renal function)
Therapies | through study completion, an average of 1 year
  Description of the therapies applied in the treatment of pathologies, report of side effects

CONTACTS AND LOCATIONS:
Overall Officials: Renato A Sinico, MD, Principal Investigator — Università degli Studi di Milano Bicocca
Locations (8):
- Italy (8):
  - ASST Lariana, Ospedale Sant' Anna, San Fermo della Battaglia, Como
  - ASST Nord Milano, Presidio Ospedaliero Bassini, Cinisello Balsamo, Milano
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - ASST Monza, Ospedale di Desio, Desio, Monza E Brianza
  - ASST Lecco, Presidio Ospedaliero Alessandro Manzoni, Lecco
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Monza, Monza
  - ASST Sette Laghi, Ospedale di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: Undecided